CLINICAL TRIAL: NCT05717348
Title: An Open-label, Multicenter, Dose-escalation and Cohort Expansion Phase 1 Clinical Study of ES014 Administered in Patients Locally Advanced or Metastatic Solid Tumours
Brief Title: A Study of ES014 in Patients With Locally Advanced or Metastatic Solid Tumours
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Elpiscience (Suzhou) Biopharma, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Elpiscience Biopharma, Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ES014-1002
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor; Locally Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: CD39; TGF-β; CD39xTGF-β
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 dose escalation (Experimental): ES014 doses will be escalated in patients with advanced solid tumors.
  Interventions: Drug: ES014
- Part 2 dose expansion (Experimental): Part 2 of the study will consist of 4 expansion cohorts at the recommended optimal biological dose determined in Part 1 dose escalation.
  Interventions: Drug: ES014

INTERVENTIONS:
Drug: ES014 — ES014 is administered via intravenous infusion, once every 14 days, every 28 days as a treatment cycle for a maximum treatment duration per patient of 2 years.

SUMMARY:
The purpose of this first-in-human, open-label, multicenter, non-randomized study designed to determine the maximum tolerated dose (MTD)/maximum administered dose (MAD), optimal biological dose (OBD), and recommended phase 2 dose (RP2D) of ES014 by evaluating the safety, tolerability, PK, pharmacodynamics, and preliminary clinical activity of ES014 administered intravenously to subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Unresectable locally advanced or metastatic solid tumour diagnosed by pathology or cytology and which meets the criteria of 1) disease progression has occurred despite receiving standard treatment and no other standard treatment is available; or 2) standard treatment has been proven to be ineffective, intolerant or considered unsuitable.

  2. Provide tumor tissue samples.

  3. At least one measurable lesion per RECIST v1.1.

  4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1. Part 1: ECOG PS 0-1. Part 2: ECOG PS 0-2.

  5. Life expectancy of at least 12 weeks.

  6. Adequate hematologic, hepatic, renal and coagulation functions per protocol.

  7. Male and female subjects of childbearing potential must be willing to completely abstain or agree to use a highly effective method of contraception.

Exclusion Criteria:

* 1. Any prior therapy targeting CD39, CD73, adenosine A2A receptor, or TGF-β.

  2. Receipt of any investigational agents or devices within 4 weeks prior to the first dose of study drug.

  3. Prior treatment with the following therapies: 1) Anticancer therapy within 30 days or 5 half-lives of the drug prior to the first dose of study drug. At least 14 days must have elapsed between the last dose of prior anticancer agent and the first dose of study drug is administered with certain exceptions. 2) A wash out of at least 2 weeks before the start of study drug for radiation to the extremities and 4 weeks for radiation to the chest, brain, or visceral organs is required.

  4. Prior allogeneic or autologous bone marrow transplantation or solid organ transplantation.

  5. Toxicity from previous anticancer treatment per protocol.

  6. Treatment with systemic immunosuppressive medications within 4 weeks prior to the first dose of study drug.

  7. Subjects who received transfusion of blood products (including platelets or red blood cells), G-CSF, GM-CSF, recombinant erythropoietin, or recombinant thrombopoietin within 14 days prior to the first dose of study treatment.

  8. Major surgery within 4 weeks prior to the first dose of study treatment.

  9. Live vaccine therapies within 4 weeks prior to the first dose of study treatment.

  10. Recent history of allergen desensitization therapy within 4 weeks prior to the first dose of study treatment.

  11. Known allergies to CHO-produced antibodies, which in the opinion of the Investigator suggests an increased potential for an adverse hypersensitivity to ES014.

  12. Invasive malignancy or history of invasive malignancy other than disease under study within the last two years per protocol.

  13. CNS metastases.

  14. Active autoimmune disease or documented history of autoimmune disease that required systemic steroids or other immunosuppressive medications per protocol.

  15. Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids or other immunosuppressive medications.

  16. Active infection requiring systemic therapy, known human immunodeficiency virus (HIV) infection, or positive test for hepatitis B active infection (HBsAg) or hepatitis C active infection (hepatitis C antibody).

  17. Current active liver or biliary disease with certain exceptions.

  18. History or evidence of cardiac abnormalities per protocol.

  19. History of bleeding tendency or a recent major bleeding event which, in the opinion of the investigator, indicates that the subject is at high risk of receiving study treatment.

  20. Pregnant or nursing females.

  21. Any known, documented, or suspected history of substance abuse that would preclude subject from participation with certain exceptions.

  22. Any other disease or clinically significant abnormality in a laboratory parameter, including serious medical or psychiatric disease/condition, that in the opinion of the investigator may compromise the safety of the subject or the integrity of the study, interfere with the subject's participation in the trial or affect the purpose of the trial.

  23. Those involved in the design and/or implementation of the study.

  24. Those deemed by the investigator to be unable to comply with the steps, limitations and requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
The frequency and severity of adverse events of ES014 | 1-3 years
  Adverse events will be assessed and assigned by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Dose Limiting Toxicity of ES014 | 1-3 years
  Evaluation of dose-limiting toxicity (DLT)

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of ES014 | 1-3 years
  Maximum observed serum concentration (Cmax) of ES014 will be measured.
Trough observed serum concentration (Ctrough) of ES014 | 1-3 years
  Trough observed serum concentration (Ctrough)of ES014 will be measured.
Area under the serum concentration time curve (AUC) of ES014 | 1-3 years
  Area under the serum concentration time curve (AUC) of ES014 will be measured.
Time to Cmax (Tmax) of ES014 | 1-3 years
  Time to Cmax (Tmax) of ES014 will be measured.
The terminal elimination half life of ES014 | 1-3 years
  The terminal elimination half-life (t 1/2) of ES014 will be measured.
The clearance of ES014 | 1-3 years
  A pharmacokinetic measurement of the volume of plasma from which ES014 is completely removed per unit time.
The volume of distribution of ES014 | 1-3 years
  The amount of of ES014 in the body divided by the plasma concentration will be measured.
The immunogenicity of ES014 | 1-3 years
  The presence and the frequency of anti-drug antibodies (ADA) against ES014 will be measured.
The antitumor activity of ES014 | 1-3 years
  Tumor response will be measured by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) by Investigator assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No